CLINICAL TRIAL: NCT04974203
Title: Saliva-based COVID-19 DNA Aptamer Test: Formative Usability and Internal Validation Study
Brief Title: Saliva-based COVID-19 DNA Aptamer Test
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Achiko AG (Industry)
Collaborators: Udayana University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2021.03.3.0102
Record Dates: First submitted 2021-07-20; First posted 2021-07-23 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Covid19
Keywords: Saliva-based test; DNA aptamer
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Patients who undertake PCR test are asked to provide saliva sample
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors are blinded to the PCR test result
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CT Value <25 (Experimental): Patients with CT value <25
  Interventions: Device: AptameX
- CT Value 25+ (Experimental): Patients with CT value of 25 or higher
  Interventions: Device: AptameX
- Negative (Experimental): Patients with negative PCR test result
  Interventions: Device: AptameX

INTERVENTIONS:
Device: AptameX — DNA aptamer-based test using patient's saliva

SUMMARY:
This study aims to conduct formative usability and internal validation of the COVID-19 rapid diagnostic test tool based on DNA aptamers, involving 200 patients to assess aspects of experimental setup, testing center, testing kit configuration, designing algorithms or workflows for clinical trials, and also assess initial accuracy by validating with the patient's PCR test results.

DETAILED DESCRIPTION:
RT-PCR has several limitations that need to be considered in its role as a COVID-19 diagnostic modality, especially in areas with limited health infrastructure. Potential diagnostic tests are needed that are capable of detecting results that are fast to read, can be carried out in service locations with limited infrastructure, and have high accuracy. The DNA Aptamers-based diagnostic test has the potential to meet these criteria, as it allows the detection of infection quickly and without invasive procedures, where the examination is only on a person's saliva.

The development of diagnostic tools must be well planned including the usability and internal validation of the tools to be studied before they can be used in clinical trial settings or diagnostic accuracy tests by involving patients in health services. This study aims to conduct formative usability and internal validation of the DNA aptamer-based COVID-19 rapid diagnostic test, involving 200 patients and also laboratory personnel to assess aspects of experimental setup, testing center, testing kit configuration, designing algorithms or workflows for testing in clinical trials, and also assess early indications of instrument accuracy by validating with the patient's PCR test data.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-59 years old
* Undertaking PCR swab test for screening, or
* In-patients undertaking PCR swab test

Exclusion Criteria:

* Unable to produce saliva
* Refusing to participate

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Hands-On-Time (HOT) | 1 month
  Total time (seconds) spent by the Operator(s) to process one test
Time-To-Result (TTR) | 1 month
  Instrument readout, from loading the cuvette in the spectrophotometer, up to recording the test as Positive / Negative
Testing Centre First-Time-Hit percentage (FTH) | 1 month
  The FTH percentage measures proportion of test kits that will be correctly processed with no single mistake, from the opening of the test kit to recording the test result.
Technician Subjective elements | 1 month
  Aspects of the workflow liked/not liked by the technicians
Patient subjective elements | 1 month
  Aspects of the workflow liked/not liked by the patient during saliva collection

SECONDARY OUTCOMES:
Sensitivity | 1 month
  The ability of a test to correctly identify those with the disease (true positive rate)
Specificity | 1 month
  The ability of the test to correctly identify those without the disease (true negative rate)
Positive Predictive Value | 1 month
  The proportions of positive results that are true positive results
Negative Predictive Value | 1 month
  The proportions of negative results that are true negative results

CONTACTS AND LOCATIONS:
Locations (1):
- Udayana University Hospital, Badung, Bali, Indonesia

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be managed by investigators only. Analyzed data or result summary will be shared to related researchers or other parties